CLINICAL TRIAL: NCT02333383
Title: A Prospective, Mono-Country, Multi-Center Study to Observe the Frequency of Extra-Axial Symptoms in Korean Ankylosing Spondylitis Patients on Adalimumab Therapy
Brief Title: Observe the Frequency of Extra-Axial Symptoms in Korean Ankylosing Spondylitis (AS) Patients
Acronym: AS PMOS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-238
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Ankylosing Spondylitis
Keywords: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score; EAMs; Adalimumab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Ankylosing Spondylitis: Adalimumab 40 mg every other week by subcutaneous (SC) injection for 52 weeks
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira; ABT-D2E7

SUMMARY:
This was a prospective mono-country, multi-center study of the frequency of extra-axial manifestations (EAMs) in Ankylosing Spondylitis (AS) participants treated with adalimumab in routine clinical practice.

DETAILED DESCRIPTION:
A baseline assessment was performed prior to the first dose of adalimumab. Participants received 40 mg of adalimumab every other week for one year. Study visits were conducted at 12, 28, 36 and 52 weeks. All participants were to have one follow-up approximately 70 days after the last dose of adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥19 years of age
* Participant has been diagnosed with ankylosing spondylitis (AS) according to the 1984 modified New York criteria for at least 3 months
* Participant has active disease defined by a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥4, despite treatment with at least 2 nonsteroidal anti-inflammatory drugs (NSAIDs) or with disease-modifying antirheumatic drugs (DMARDs) for more than 3 months based on Korea AS reimbursement guideline
* Participant is eligible for adalimumab in daily rheumatologic practice
* Participant must provide written authorization form to use personal and/or health data prior to the entry into the study

Exclusion Criteria:

* Female participants who are pregnant or breastfeeding
* Participants who are contraindicated to any anti-tumor necrosis factor (TNF) agent
* Participant is enrolled in other clinical trials

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2014-12-31; Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EunJung Gu, Study Director — AbbVie Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intention-to-Treat (ITT) population: Participants who received at least one dose of adalimumab and had extra-axial manifestations (EAMs) assessed at baseline
Period: Overall Study
Arm/Group | Participants With Ankylosing Spondylitis
Started | 201
Completed | 160
Not Completed | 41
Not completed — Adalimumab discontinuation | 21
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 3
Not completed — Transfer to another hospital | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population: Participants who received at least one dose of adalimumab and had extra-axial manifestations (EAM) assessed at baseline
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.84 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 201
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Extra-Axial Manifestations (EAMs) of Interest
Description: The baseline assessment was performed prior to the first dose of adalimumab. The presence of peripheral arthritis (arthritis affecting shoulders, elbows, wrists, hands, knees, ankles, feet), enthesitis (inflammation of the areas where ligaments or tendons insert into bone) and dactylitis (inflammation of finger and/or toe joints) was noted. Peripheral arthritis was defined as ≥1 swollen joint on the Swollen Joint Count scale (SJC; range, 0 to 44, excluding hip joints). Enthesitis was defined as at least one inflamed enthesis in the Maastricht Ankylosing Spondylitis Enthesitis Score (MASES, 0 to 13, with higher scores representing more severe disease) or of the plantar fascia of the foot. Dactylitis was measured by a simple count of dactylitic digits.
Time Frame: Baseline
Population: Intention-to-Treat (ITT) population: Participants who received at least one dose of adalimumab and had extra-axial manifestations (EAMs) assessed at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 201
Percentage of participants
  Enthesitis | 46.27 [39.23 to 53.42]
  Peripheral arthritis | 33.33 [26.86 to 40.31]
  Dactylitis | 2.99 [1.10 to 6.38]

2. Secondary Outcome: Proportion of Participants Achieving a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response
Description: The Bath Ankylosing Spondylitis (AS) Disease Activity Index assesses disease activity by asking the participant to answer 6 questions (each on a 10 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity. BASDAI 50 is a 50% improvement from baseline in BASDAI score.
Time Frame: Baseline, Week 12, Week 28, Week 36, Week 52
Population: Intention-to-Treat (ITT) population: Participants with available data who received at least one dose of adalimumab and had extra-axial manifestations (EAMs) assessed at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 189
Participants
  Week 12 | 142
  Week 28: number analyzed (Participants) | 155
  Week 28 | 128
  Week 36: number analyzed (Participants) | 162
  Week 36 | 142
  Week 52: number analyzed (Participants) | 144
  Week 52 | 130

3. Secondary Outcome: Mean Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) in Participants With Enthesitis at Baseline
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Each domain was graded for the presence (1) or absence (0) of tenderness yielding total MASES ranging from 0 (0 sites with tenderness) to 13 (worst possible score; 13 sites with tenderness). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12, Week 28, Week 36, Week 52
Population: Intention-to-Treat (ITT) population: Participants with available data who received at least one dose of adalimumab and had enthesitis at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 86
units on a scale
  Week 12: number analyzed (Participants) | 84
  Week 12 | -1.85 (2.50)
  Week 28: number analyzed (Participants) | 72
  Week 28 | -2.31 (2.03)
  Week 36: number analyzed (Participants) | 71
  Week 36 | -2.31 (1.78)
  Week 52: number analyzed (Participants) | 68
  Week 52 | -2.50 (1.90)

4. Secondary Outcome: Proportion of Participants With Enthesitis of the Plantar Fascia
Description: The plantar fascia is a ligament that runs along the bottom of each foot. The percentage of participants who had enthesitis of the plantar fascia was documented at each study visit.
Time Frame: Baseline, Week 12, Week 28, Week 36, Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 201
Participants
  Baseline | 19
  Week 12: number analyzed (Participants) | 193
  Week 12 | 10
  Week 28: number analyzed (Participants) | 173
  Week 28 | 2
  Week 36: number analyzed (Participants) | 169
  Week 36 | 4
  Week 52: number analyzed (Participants) | 160
  Week 52 | 7

5. Secondary Outcome: Mean Change in Dactylitis Score in Participants With Dactylitis at Baseline
Description: Assessment of the presence or absence of dactylitis (inflammation of finger and/or toe joints) as well as grading of tenderness and swelling in all 20 of the participants' digits was performed. Tenderness at each site was quantified from absent to severe. Swelling was quantified from mild to severe. Total Dactylitis Assessment scores ranged from 0 (no digits with dactylitis) to 20 (worst possible score; 20 digits with dactylitis). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12, Week 28, Week 36, Week 52
Population: Intention-to-Treat (ITT) population: Participants with available data who received at least one dose of adalimumab and had dactylitis at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 6
units on a scale
  Week 12 | -3.83 (3.66)
  Week 28: number analyzed (Participants) | 5
  Week 28 | -4.40 (3.78)
  Week 36: number analyzed (Participants) | 4
  Week 36 | -5.00 (4.08)
  Week 52: number analyzed (Participants) | 4
  Week 52 | -5.00 (4.08)

6. Secondary Outcome: Mean Change in Tender Joint Counts (TJC) in Participants With Peripheral Arthritis (≥1 Swollen Joint) at Baseline
Description: Forty-six joints were assessed for tenderness by physical examination. Tenderness of each joint was classified as present (1) or absent (0), for a total possible TJC score of 0 (0 joints with tenderness) to 46 (worst possible score/46 joints with tenderness). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12, Week 28, Week 36, Week 52
Population: Intention-to-Treat (ITT) population: Participants with available data who received at least one dose of adalimumab and had peripheral arthritis (≥1 swollen joint) at baseline
Measure: Mean (Standard Deviation); unit: Tender joint counts
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 67
Tender joint counts
  Week 12: number analyzed (Participants) | 66
  Week 12 | -1.82 (3.43)
  Week 28: number analyzed (Participants) | 56
  Week 28 | -2.05 (3.03)
  Week 36: number analyzed (Participants) | 53
  Week 36 | -2.38 (3.13)
  Week 52: number analyzed (Participants) | 50
  Week 52 | -2.60 (2.87)

7. Secondary Outcome: Mean Change in Change in Swollen Joint Counts (SJC) in Participants With Peripheral Arthritis (≥1 Swollen Joint) at Baseline
Description: Forty-four joints, excluding hip joints, were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score SJC of 0 (0 joints with swelling) to 44 (worst possible score/44 joints with swelling). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 12, Week 28, Week 36, Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Swollen joint counts
Arm/Group | Participants With Ankylosing Spondylitis
Number analyzed (Participants) | 67
Swollen joint counts
  Week 12: number analyzed (Participants) | 66
  Week 12 | -1.80 (2.25)
  Week 28: number analyzed (Participants) | 56
  Week 28 | -1.98 (2.79)
  Week 36: number analyzed (Participants) | 53
  Week 36 | -2.04 (2.86)
  Week 52: number analyzed (Participants) | 50
  Week 52 | -2.40 (2.30)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 70 days after the last dose of study drug (up to 62 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Participants With Ankylosing Spondylitis
All-Cause Mortality (participants affected / at risk) | 0/201
Serious Adverse Events (participants affected / at risk) | 8/201
Other Adverse Events (participants affected / at risk) | 18/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Ankylosing Spondylitis (N=201)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Ankylosing Spondylitis (N=201)
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Cellulitis (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Uveitis (Eye disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT02333383/Prot_SAP_000.pdf